CLINICAL TRIAL: NCT03527108
Title: A Phase 2 Study of Nivolumab Plus Ramucirumab in Patients With Recurrent, Advanced, Metastatic Non-Small Cell Lung Carcinoma
Brief Title: Nivolumab Plus Ramucirumab in Patients With Recurrent, Advanced, Metastatic NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-189; TH-189 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Immunotherapy; Ant-angiogenic therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with prior IO therapy (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ramucirumab

INTERVENTIONS:
Drug: Nivolumab — The treatment will be given on a 28-day cycle, with doses of nivolumab and ramucirumab given on days 1 and 15. The dose of nivolumab will be fixed at 240 mg. Nivolumab should be administered first, followed by premedication, and then ramucirumab. Ramucirumab should be administered approximately 30 minutes after premedication
Drug: Ramucirumab — The treatment will be given on a 28-day cycle, with doses of nivolumab and ramucirumab given on days 1 and 15. The dose of ramucirumab will depend upon the patient weight as noted below. Nivolumab should be administered first, followed by premedication, and then ramucirumab. Ramucirumab should be administered approximately 30 minutes after premedication

SUMMARY:
The study will enroll patients with prior IO therapy (alone or in combination with chemotherapy or in combination with other IO agents) regardless of the PD-L1 level, into a non-randomized combination trial, with primary endpoint of disease control rate.

DETAILED DESCRIPTION:
Immunotherapeutic treatment with check-point inhibitors has increased survival in patients with advanced non-small cell lung cancer (NSCLC) that does not have any mutation to be targeted. However, the concept that tumors evade immune surveillance through a variety of mechanisms, and that activating the immune system can lead to tumor regression in a variety of tumor types has been known for decades. Thus, this study combines the effects to blocking 2 different pathways- inhibition of PD-1 pathway and angiogenic pathway via inhibition of VEGR signaling to improve survival as blocking each pathway individually has demonstrated a modest increment. There has been no study using nivolumab in combination with a VEGFR2 inhibitor, a drug which has both anti-angiogenic and pleotropic immunomodulatory effects and may synergize with the effect of an anti-PD-1 agent, in solid tumors. Activating the anti-tumor effects of T cells by utilizing multiple pathways of both nivolumab and ramucirumab is an endeavor which merits investigation.

Thus, the study investigates the synergistic effect of targeted anti-antitumor activity of immune checkpoint inhibitor nivolumab and immune-suppressive activity of VEGF-inhibitor ramicirumab expecting a favorable overall survival in NSCLC patients, with the additional benefit of tolerable toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed, refractory or recurrent, advanced non-small cell lung carcinoma regardless of histology.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 as described in detail in section 11.0
3. Patients must have completed one line of prior therapy in both cohorts. For participation in the Cohort A, they must have completed at least 4 cycles of platinum doublet therapy. For participation in Cohort B, they must have received PD-1, PD-L1 and/or CTLA-4 immunotherapy, alone or in combination with chemotherapy or in combination with other IO agents. Treatment on this protocol may begin as long as the patient has recovered from toxicities of prior therapy at the discretion of the treating physician. A washout period of at least 2 weeks is required prior to starting on this trial.
4. Patients with recurrent disease who had received adjuvant or neoadjuvant therapy or chemoradiotherapy for locally advanced disease if their disease has progressed up to 6 months after completion of adjuvant or neoadjuvant platinum-based therapy, or if their disease has progressed more than 6 months after therapy and during or after a subsequent platinum-based chemotherapy regimen
5. Patients with molecular targets (EGFR, ALK, ROS1) who have progressed on targeted agents and are not eligible for other treatments or trials specific for this population are allowed.
6. Age > 18 years.
7. ECOG performance status 0 or 1
8. Patients must have normal organ and marrow function as defined below. Patients should be able to maintain ANC levels without the need for G-CSF transfusion. If blood transfusion is performed for achieving hemoglobin levels, the levels should stay at ≥ 9.0 mg/ml for at least a week after transfusion.

   Absolute neutrophil count > 1,500/mcL Hemoglobin ≥ 9.0 mg/ml Platelets > 100,000/mcL Total bilirubin ≤1.5 X institutional upper limit of normal (ULN) AST/ALT (SGOT/SGPT) < 3 times institutional normal limits, or up to 5 times institutional normal limits if the patient has liver metastases Creatinine OR Creatinine clearance ≤1.5 X ULN, OR > 40 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal as per Cockcroft-Gault formula International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) <1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). If receiving warfarin, the patient must have an INR ≤3.0. For heparin and LMWH there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
10. Ability to understand and willingness to sign a written informed consent and HIPAA consent document
11. A core tumor biopsy obtained after progression on the last treatment must be available at study entry for the study. The biopsy sample must not be more than 90 days old at the time of registration and the sample must be adequate for analyses. If the sample is not adequate patient must agree to provide a fresh biopsy specimen before the start of treatment. Any available archival tissue will also be collected.
12. The patient's urinary protein must be ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).
13. Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication.
14. Female subjects of childbearing potential and male subjects must be willing to use an effective method of contraception - Contraception, for the course of the study through 150 days after the last dose of study medication.
15. Male patients who have women of child bearing potential (WOCBP) partners must agree to use effective method of contraception - Contraception, for the course of the study through 210 days after the last dose of study medication.
16. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Patients who have not recovered from their most recent chemotherapy or radiotherapy prior to entering the study at the discretion of investigators. Patients may not be currently receiving any other investigational agents or immunomodulatory agents (e.g. ipilimumab). Patients treated with prior PD-1 or PD-L1 directed therapies are ineligible Cohort A.
2. Prior ramucirumab treatment
3. The patient has experienced any Grade 3-4 GI bleeding within 3 months prior to first dose of protocol therapy.
4. The patient has a history of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy.
5. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
6. The patient has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy.
7. The patient has uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
8. The patient with history of hemoptysis (defined as bright red blood or ≥ 1/2 teaspoon) within 2 months prior to first dose of protocol therapy or with radiographic evidence of intra-tumor cavitation or has radiologically documented evidence of major blood vessel invasion or encasement by cancer.
9. The patient has a serious or non-healing wound, ulcer, or bone fracture (as per physician's discretion) within 28 days prior to first dose of protocol therapy.
10. The patient has a prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation.
11. The patient has undergone major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
12. The patient is receiving chronic antiplatelet therapy other than aspirin, including nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted. Occasional use of NSAIDS is allowed (occasional use would constitute daily use for less than a week; treating physician discretion is permitted to differentiate between occasional Vs chronic use).
13. Patients who have not recovered from adverse events due to agents administered earlier except neuropathy and alopecia. Physician's discretion is allowed to decide which unresolved adverse events from previous therapy (for NSCLC) prohibit patient participation in this study.
14. Patients with active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Hormone replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Patients requiring more than 10mg prednisolone (or its equivalent) per day are excluded.
16. Patients with untreated symptomatic brain metastases are excluded. Patients with treated brain metastases will be allowed if brain imaging obtained within 28 days of trial enrollment reveals stable disease. Patients with small (<5mm) asymptomatic brain metastasis are allowed to enroll.
17. Patients with interstitial lung disease or active, noninfectious pneumonitis. Patients with active tuberculosis infection are excluded.
18. Patient who have received a live vaccine within 30 days prior to Cycle1 Day 1.
19. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (significant), cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
20. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
21. Known history of chronic hepatitis B virus infection or chronic hepatitis C virus indicating chronic infection that is not cured.
22. Subjects with previous malignancies (except non-melanoma skin cancers, and in situ cancers such as the following: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
23. Pregnant or breast-feeding.
24. Patients with prior grades 3 and 4 immune related adverse effects as a result of prior therapy with a checkpoint inhibitor are excluded

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) in IO experienced patients.treated with nivolumab and ramucirumab combination therapy | 12 months
  DCR is defined as number of patients with stable disease, complete or partial response as determined by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 12 months
  ORR is defined as the number of patients with partial response or complete response as determined by RECIST 1.1 criteria
Progression free survival (PFS) at 6 months | 12 months
  Number of patients with progression free survival (PFS). 1. PFS is defined as the length of time from the start of treatment to time of disease progression or death, whichever occurs first, as determined by RECIST 1.1 criteria
Number of patients with treatment related toxicities in IO naive patients treated with nivolumab and ramucirumab combination therapy | 12 months
  Toxicity is determined by NCI Common Toxicity Criteria for Adverse Events (CTCAE) v4.03
Overall survival in IO experienced patients treated with nivolumab and ramucirumab combination. | 60 months
  Defined by the number of patients alive at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Borghaei, DO, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - NYU Langone, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania